CLINICAL TRIAL: NCT02116101
Title: Evaluation of the Effect of Momchilovtsi Yogurt on Intestinal Health and Blood Lipid Adjustment in Human Subjects
Brief Title: Intestinal Health and Blood Lipid Adjustment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bright Dairy & Food Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 12-SC-11-BRD-001
Record Dates: First submitted 2014-04-12; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Constipation
Keywords: Intestinal Health; Prebiotics; Blood Lipid
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bright Momchilovtsi yogurt (Active Comparator): Bright Momchilovtsi yogurt Contains 1×106cfu/g prebiotics including Lactobacillus bulgaricus and Streptococcus thermophilus
  Interventions: Dietary Supplement: Bright Momchilovtsi Yogurt
- Bright Dairy Beverage (Placebo Comparator): Dairy beverage product without prebiotics
  Interventions: Dietary Supplement: Bright Dairy Beverage

INTERVENTIONS:
Dietary Supplement: Bright Momchilovtsi Yogurt — Oral consumption of Bright Momchilovtis Yogurt containing 1×106cfu/g prebiotics including Lactobacillus bulgaricus and Streptococcus thermophilus
  Dosage: 110g at a time, twice per day at 10 am and 4 pm. Duration: 7 weeks (March 10, 2013 - April 27, 2013) The active study product has similar package and taste as the placebo.
  Arms: Bright Momchilovtsi yogurt
Dietary Supplement: Bright Dairy Beverage — Oral consumption of Bright Dairy Beverage Dosage: 110g at a time, twice per day at 10 am and 4 pm. Duration: 7 weeks (March 10, 2013 - April 27, 2013) The active study product has similar package and taste as the placebo.
  Arms: Bright Dairy Beverage

SUMMARY:
This was a randomized, double-blind, single-center, placebo-controlled, two-arm study. The objectives of this study were to evaluate the effect of Momchilovtsi yogurt on:

1. Improving intestinal digestion and bowl movement;
2. Adjusting blood total Cholesterol and Triglycerides levels;
3. Adjusting microbiological flora (Clostridium perfringens bacteria, Lactobacillus and Bifidobacterium) in gastrointestinal tract;
4. Adjusting short chain fatty acids (acetic acid, propionic acid, butyric acid) in in gastrointestinal tract.

DETAILED DESCRIPTION:
1. Quality control of the study:

   1.1 Study monitoring and source data verification:

   Monitoring was done according to the monitoring plan by a representative of the investigator, who checked the case report forms for completeness and clarity, and cross-checked them with source documents. In addition to the monitoring visits, frequent communications (letter, telephone, fax, e-mail), by the study monitor ensured that the investigation was conducted according to protocol design and regulatory requirements. Study close-out was performed by the study monitor upon closure of the study.

   1.2 On-site audits:

   Domestic and foreign regulatory authorities, the Institutional Review Board, and an auditor authorized by the sponsor may request access to all source documents, case report forms, and other study documentation for on-site audit or inspection. Direct access to these documents was guaranteed by the investigator, who must provide support at all times for these activities. Medical records and other study documents may be copied during audit or inspection provided that subject names are obliterated on the copies to ensure confidentiality.

   1.3 Documentation:

   A case report form was provided for each subject.

   All protocol-required information collected during the study was entered by the investigator, or designated representative, in the case report form. Details of case report form completion and correction were explained to the investigator.

   The investigator, or designated representative, should complete the case report form pages as soon as possible after information is collected, preferably on the same day that a study patient is seen for an examination, treatment, or any other study procedure. Any outstanding entries must be completed immediately after the final examination. An explanation should be given for all missing data.

   A source data location list was prepared prior to study initiation. This list was filed in both the trial master file and the investigator study file and updated as necessary.

   The completed case report forms were reviewed and signed by the investigator named in the clinical study protocol or by a designated sub investigator.

   The sponsor would retain the original of all completed case report forms. The principal investigator kept the copies of all completed case report forms for 25 years after the trial based on Good Clinical Practice requirements.
2. Quality assurance of study products:

   All products used in this study were manufactured and provided by Bright Dairy & Food Co., Ltd. The quality test of study products was conducted by Shanghai dairy products quality supervision and inspection station. The study products were stored at the study site and assigned to the subjects by the investigator. The amount of products received and assigned were filed on product distribution list by the investigator. The study products were not allowed to be given to anyone who didn't participated in the study. No sales of unassigned products was allowed. After the completion of the study, the unassigned products need to be returned to Bright Dairy & Food Co., Ltd.

   The products were labeled with study code. A master participation list was completed which identifies each patient full name and unique identification number. The identity of the specific product was blind to patients, support staff and investigators. The unmasking occurred to the investigators and statistical analyses team only after completion of statistical analyses.
3. Data management:

   Study data were recorded on Case Report Forms (CRFs) and then entered into saved in the form of Excel files. Data was double entered and cross-validated.
4. Management of subject withdrawal:

   A number of 120 subjects were enrolled in the study.

   Subjects may be withdrawn from the study for the following reasons:
   * At their own request or at the request of their legally authorized representative,
   * If, in the investigator's opinion, continuation in the study would be detrimental to the patient's well-being,
   * If they are lost to follow-up.

   In all cases, the reason for and date of withdrawal must be recorded in the Exit Form and in the subject's medical records and the sponsor's representative must be notified within 5 days. The subject must be followed up to establish whether the reason was an adverse event, and, if so, this must be reported in accordance with the procedure of an adverse event (described bellow). The investigator must make every effort to contact subject lost to follow-up. Attempts to contact such subject must be documented in the subject's records (e.g., dates and times of attempted telephone contact).

   Investigator must be notified of all serious or unexpected adverse events within 48 hours. Notification does not depend on whether there is a connection to the study formula or not. All adverse events must be documented on the appropriate pages of the case report forms.
5. Statistical analysis plan:

Analysis was performed for the intent-to-treat population.

Chi-square test was used comparison between study groups for categorical data. For continuous outcomes, t-test was used for between-group comparison, paired t-test was used for pre-post comparison within each study group.3. Non-parametric methods were used for non-normal data, data with unequal variances. The analysis was completed using the statistical package SPSS17.0.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 30-60 years;
* Abnormal blood lipids level;
* Have aperiodic or occasional gastrointestinal symptom (gastrointestinal tympanites, abnormal borborygmus, heavy feeling after meal, celiodynia, abdominal pain);
* Slow power of intestinal tract or irregular intestinal moving (abnormal feces solidity, decreased feces quantity, e.g. defecate every 2-3 days or defecate less than 3 times a week)

Exclusion Criteria:

* Diagnosed as chronic constipation;
* Receiving treatment for gastrointestinal symptoms;
* Lactose Intolerance;
* In use of analgesic such as aspirin or Panadol, etc;
* Have had laxatives or other substance that will enhance digestion within 2 weeks before the study begins;
* Have had dairy products or other food containing probiotics within 10 days before the study begins;
* Have diarrhea currently;

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in health status of the intestinal tract at Day 49 | Day 0, 49
  Weekly stool frequency (>6; 4-6; 1-3; 0)
  Ratio of unopened defecation times vs. total defecation times (0; 1/4; 1/3; ≥1/2)
  Duration of defecation (<5 min; 5-15 min; 16-30 min; ≥30 min)
  Defecation condition (normal perception; straining/uncomfortableness at stool; obvious straining/uncomfortableness or difficulty at stool, little feces quantity; frequent symptom of celialgia or calor at anus, which affect defecation)

SECONDARY OUTCOMES:
Blood total cholesterol level (mmol/L) | Baseline (day 0), day 49
Blood triglycerides level (mmol/L) | Baseline (day 0), day 49
Fecal bacterium counts | Baseline (day 0), day 49
  Fecal bacterium including Clostridium perfringens bacteria, Lactobacillus and Bifidobacterium
Fecal short chain fatty acids (%) | Baseline (day 0), day 49
  Acetic acid, propionic acid, butyric acid
Score of digestive system (score 0-10) | Day 0, 7, 14, 21, 28, 35, 42, 49
  Abdominal distention, abdominal pain, gastric distention, heavy stomach, loss of appetite, belching
Satisfaction with Defecation Habit | Day 0, 7, 14, 21, 28, 35, 42, 49
  Satisfied / Unsatisfied on: Defecation frequency, defecation duration , stool characteristic, and defecation habit

CONTACTS AND LOCATIONS:
Overall Officials: Donglian Cai, MD, Principal Investigator — Department of Nutrition, The Second Military Medical University Affilated Changhai Hospital